CLINICAL TRIAL: NCT00556452
Title: Phase I/II Study of Myeloablative Allogeneic Stem Cell Transplantation for Aggressive Hematologic Malignancies Using Clofarabine and Busulfan x 4 (Clo/BU4) Regimen
Brief Title: Study of Stem Cell Transplantation for Hematologic Malignancies Using Clofarabine and Busulfan Regimen
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2007.055
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Leukemia; Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Multiple Myeloma; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia; Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma; Myelodysplastic Syndromes | interventions — Clofarabine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clo/BU4 (Experimental): Study will start at the 2nd dose level of three Clofarabine levels, in combination with Busulfan. The Clofarabine level that each subsequent patient is treated at is determined by a method using continual reassessment.
  After pre-conditioning, subjects will receive a peripheral blood stem cell transplant.
  Interventions: Drug: Clofarabine/Busulfan x 4; Procedure: Peripheral blood stem cell transplant; Radiation: Total Lymphoid Irradiation

INTERVENTIONS:
Drug: Clofarabine/Busulfan x 4 — Clofarabine IV (dose levels)
  * 1st dose level: 20 mg/m2/day x 5 days
  * 2nd dose level: 30 mg/m2/day x 5 days
  * 3rd dose level: 40 mg/m2/day x 5 days
  Busulfan IV 3.2 mg/kg daily x 4 days
Procedure: Peripheral blood stem cell transplant — Peripheral blood stem cell transplant, after pre-conditioning drug treatment
Radiation: Total Lymphoid Irradiation — Total Lymphoid Irradiation (TLI) of 4 Gy, if cord blood transplant

SUMMARY:
The goals of the study are (Phase I) to determine the appropriate dose for Clofarabine with Busulfan as a full-intensity conditioning (Clo/BU4 regimen) prior to transplant and then (Phase II) to investigate the safety and effectiveness of this regimen as a conditioning for stem cell transplant in the treatment of aggressive hematologic malignancies in subjects where more conventional approaches are failing.

DETAILED DESCRIPTION:
Transplants with stem cells collected from the blood of an unrelated donor (allo-HSCT) are being used more commonly for many blood cancers which are not curable with more conventional methods of chemotherapy. Although allo-HSCT has great potential, there are still high risks due to infections, graft-versus-host disease (GVHD), where the donor's cells attack the recipient's tissues as foreign, and due to toxic effects of the chemotherapy drugs given to prepare (or condition) the recipient's bone marrow for transplant.

As a reduced intensity conditioning, a combination of Fludarabine and a lower dose of Busulfan (Flu/BU2) is one of the most popular regimens. Among full-intensity regimens, a combination of Fludarabine and standard-dose Busulfan (Flu/BU4) has been investigated recently and shown to be very well tolerated.

Clofarabine, similar to Fludarabine, is known to have a stronger anti-tumor effect than Fludarabine and has shown promise in treating aggressive acute leukemias. In addition, evidence is that it is well-tolerated with manageable side effects especially in older subjects. Thus replacing Fludarabine with Clofarabine in a full-intensity transplant regimen, Clo/BU4 may provide a regimen with increased anti-tumor activity without adding significant risks of toxicity.

The goals of the study are (Phase I) to determine the appropriate dose for Clofarabine with Busulfan as a full-intensity regimen (Clo/BU4) and then (Phase II) to investigate the safety and effectiveness of this regimen as a conditioning for HSCT in the treatment for aggressive hematologic malignancies, in subjects where more conventional approaches are failing.

ELIGIBILITY:
Inclusion Criteria:

Disease Criteria

* Acute leukemia or chronic myelogenous leukemia in blastic crisis or accelerated phase, not in remission at the time of transplant
* Myelodysplastic syndrome, with more than 5% blasts in bone marrow at the time of transplant
* Hodgkin and Non-Hodgkin Lymphomas: Not in CR in PET scan or CT scan before transplant, or relapsed within 1 year from previous remission
* CLL not in remission
* Multiple Myeloma, not in remission
* Suitable donor available (related or unrelated)

Age, Organ Function Criteria

* Age: ≤ 70 years
* Cardiac: LV Ejection Fraction ≥ 40% by MUGA or Echocardiogram
* Pulmonary: FEV1 and FVC ≥ 40% predicted, and DLCO (corrected for hemoglobin) ≥ 40% of predicted
* Renal: Adult population: serum creatinine ≤ 1.0 mg/dL (if serum creatinine > 1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be > 60 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation)
* Renal: Pediatric population: serum creatinine clearance ≥ 90 ml/min/1.73 m2 as calculated by the Schwartz formula for estimated GFR
* Hepatic: serum total bilirubin ≤ 2.0 mg/dl and AST / ALT ≤ ULN x 4
* Performance status: Karnofsky ≥ 70%

Exclusion Criteria:

* Other active life-threatening cancer requiring treatment other than allo-HSCT
* HIV1 or HIV2 positive
* Uncontrolled medical or psychiatric disorder
* Uncontrolled viral or fungal infection
* Active CNS leukemia
* Non-compliant to medications
* No appropriate caregivers identified

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-10; Primary Completion 2011-06 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Magenau, M.D., Principal Investigator — University of Michigan, Department of Internal Medicine, Blood and Marrow Transplant Program
Locations (1):
- University of Michigan, Department of Internal Medicine, Blood and Marrow Transplant Program, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Magenau J, Tobai H, Pawarode A, Braun T, Peres E, Reddy P, Kitko C, Choi S, Yanik G, Frame D, Harris A, Erba H, Kujawski L, Elenitoba-Johnson K, Sanks J, Jones D, Paczesny S, Ferrara J, Levine J, Mineishi S. Clofarabine and busulfan conditioning facilitates engraftment and provides significant antitumor activity in nonremission hematologic malignancies. Blood. 2011 Oct 13;118(15):4258-64. doi: 10.1182/blood-2011-06-358010. Epub 2011 Aug 12. PMID 21841163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with relapsed or refractory hematologic malignancies not in remission received unmanipulated HSCT with CloBu4 conditioning from October 2007 to November 2009 at the University of Michigan. Patients received a clofarabine dose of 20mg/m^2, 30 mg/m^2 or 40 mg/m^2.
Groups:
- Clo/BU4 20mg/m^2: Clofarabine/Busulfan x 4 : Clofarabine IV 20 mg/m^2/day x 5 days
  Busulfan IV 3.2 mg/kg daily x 4 days
  Peripheral blood stem cell transplant : Peripheral blood stem cell transplant, after pre-conditioning drug treatment.
- Clo/BU4 30mg/m^2: Clofarabine/Busulfan x 4 : Clofarabine IV 30 mg/m^2/day x 5 days
  Busulfan IV 3.2 mg/kg daily x 4 days
  Peripheral blood stem cell transplant : Peripheral blood stem cell transplant, after pre-conditioning drug treatment.
- Clo/BU4 40mg/m^2: Clofarabine/Busulfan x 4 : Clofarabine IV 40 mg/m^2/day x 5 days
  Busulfan IV 3.2 mg/kg daily x 4 days
  Peripheral blood stem cell transplant : Peripheral blood stem cell transplant, after pre-conditioning drug treatment.
Period: Overall Study
Arm/Group | Clo/BU4 20mg/m^2 | Clo/BU4 30mg/m^2 | Clo/BU4 40mg/m^2
Started | 6 | 21 | 19
Completed | 6 | 21 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Experimental: Clo/BU4
Groups:
- Total: Total of all reporting groups
Arm/Group | Clo/BU4 20mg/m^2 | Clo/BU4 30mg/m^2 | Clo/BU4 40mg/m^2 | Total
Number analyzed (Participants) | 6 | 21 | 19 | 46
Age, Continuous [Median (Full Range); unit: years] | 48.5 [14 to 61] | 54 [18 to 68] | 51 [1 to 67] | 53 [1 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11 | 22
  Male | 4 | 12 | 8 | 24
Region of Enrollment [Number; unit: participants]
  United States | 6 | 21 | 19 | 46
Disease [Number; unit: participants] — The number of patients with each disease type.
  participants
    Acute Myeloid Leukemia (AML) | 4 | 13 | 14 | 31
    Chronic Myeloid Leukemia (CML) | 1 | 1 | 0 | 2
    Acute Lymphoblastic Leukemia (ALL) | 1 | 1 | 2 | 4
    Chronic Lymphocytic Leukemia (CLL) | 0 | 3 | 1 | 4
    Non-Hodgkin Lymphoma (NHL) | 0 | 2 | 1 | 3
    Myelodysplastic Syndromes (MDS) | 0 | 0 | 1 | 1
    Multiple Myeloma (MM) | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Regimen Related Toxicities
Description: The incidence of non-hematological toxicities (Common Terminology Criteria for Adverse Events (CTCAE) 3.0) from initiation of conditioning to Day + 30 or toxicities after day +30, possibly, probably or definitely related to conditioning for all patients treated with Clofarabine (independent of dose level).
Time Frame: two years
Measure: Number; unit: toxicities
Groups:
- Clo/Bu4: Experimental: Clo/BU4
Arm/Group | Clo/Bu4
Number analyzed (Participants) | 46
toxicities
  Liver | 56
  Gastrointestinal | 70
  Genito-Urinary | 4
  Cardiopulmonary | 10
  Neurologic | 8
  Skin | 11
  Other | 3

2. Primary Outcome: One-year Overall Survival Rate for AML
Description: Percent Overall Survival (OS) for at one year for subjects with Acute Myeloid Leukemia (AML).
Time Frame: 1 year
Population: Patients with Acute Myeloid Leukemia (AML)
Measure: Number (95% Confidence Interval); unit: percent overall survival
Groups:
- Clo/BU4: Study will start at the 2nd dose level of three Clofarabine levels, in combination with Busulfan. The Clofarabine level that each subsequent patient is treated at is determined by a method using continual reassessment.
  After pre-conditioning, subjects will receive a peripheral blood stem cell transplant.
  Total Lymphoid Irradiation : Total Lymphoid Irradiation (TLI) of 4 Gy, if cord blood transplant
  Clofarabine/Busulfan x 4 : Clofarabine IV (dose levels)
  * 1st dose level: 20 mg/m2/day x 5 days
  * 2nd dose level: 30 mg/m2/day x 5 days
  * 3rd dose level: 40 mg/m2/day x 5 days
  Busulfan IV 3.2 mg/kg daily x 4 days
  Peripheral blood stem cell transplant : Peripheral blood stem cell transplant, after pre-conditioning drug treatment
Arm/Group | Clo/BU4
Number analyzed (Participants) | 31
percent overall survival | 48 [34 to 70]

3. Secondary Outcome: Two-year Overall Survival for All Cases.
Description: Percent Overall Survival (OS) at two years for all patients.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percent overall survival
Arm/Group | Clo/BU4
Number analyzed (Participants) | 46
percent overall survival | 28 [17 to 45]

4. Secondary Outcome: Five Year Overall Survival for All Cases
Description: The number of patients alive at 5 years
Time Frame: five years
Measure: Count of Participants; unit: Participants
Arm/Group | Clo/BU4
Number analyzed (Participants) | 46
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse events occurring following study registration, but prior to beginning transplant therapy will not be reported. Post transplant, adverse events will be reported through day 100.
Description: Adverse events were analyzed for all patients that received Clofarabine, and not by Clofarabine dose received. All patients received the same study drug, Clofarabine.
Arm/Group | Clo/Bu4
Serious Adverse Events (participants affected / at risk) | 23/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clo/Bu4 (N=46)
Ascites (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Hypoxia/Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Fever (General disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Vascular Access Complication (Vascular disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Atrial Fibrilation (Cardiac disorders) | 1
Bladder Hemmorhage (Vascular disorders) | 1
Blood Disorder (Blood and lymphatic system disorders) | 1
Death (General disorders) | 1
Disease Progression (Investigations) | 1
Dizziness (Nervous system disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Graft Versus Host Disease (Immune system disorders) | 2
Infection (Infections and infestations) | 7
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Portal Hypertension (Vascular disorders) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clo/Bu4 (N=46)
Transaminitis* (Hepatobiliary disorders) | 43
Hyperbilirubiniemia (Hepatobiliary disorders) | 8
Mucositis (Gastrointestinal disorders) | 31
Nausea/Vomiting (Gastrointestinal disorders) | 25
Diarrhea (Gastrointestinal disorders) | 10
Abdominal Pain (Gastrointestinal disorders) | 5
Creatinine elevation (Renal and urinary disorders) | 3
Headache (Nervous system disorders) | 4
Confusion (Nervous system disorders) | 1
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 2
Hypotention (General disorders) | 2
Veno-Occlusive Disease (Vascular disorders) | 2
Ascites (Gastrointestinal disorders) | 3
Hypertension (Cardiac disorders) | 3
Hemorragic Cystitis (Renal and urinary disorders) | 1
Arrythmia (Cardiac disorders) | 1
Hypersensitivity (General disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6
Syncope (Nervous system disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Fracture (Musculoskeletal and connective tissue disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 21
Deep Vein Thrombosis (Vascular disorders) | 2
Cholycytitis (Hepatobiliary disorders) | 1
Cirrhosis (Hepatobiliary disorders) | 1
Siezure (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No